CLINICAL TRIAL: NCT00749853
Title: Prospective, Randomized Open Trial to Evaluate the Efficacy of an Ovarian Stimulation Protocol Based on FSH Receptor Genotype
Brief Title: Efficacy of Ovarian Stimulation Based on FSHR Genotype Status
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: PI left the institution
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Clemens Tempfer, Prof. Clemens Tempfer, MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ufktem1
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Sterility
Keywords: ovarian stimulation; FSH; genotyping; polymorphism
MeSH Terms: conditions — Infertility | interventions — Follicle Stimulating Hormone; Buserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Pituitary down-regulation will be achieved using buserelin (Suprefact®, Hoechst, Frankfurt, Germany) at a fixed daily dose of 200 mg s.c., according to a long agonist protocol, starting on day 2 of the normal menstrual cycle. Treatment with r-hFSH (Gonal-F®, Serono Austria GmbH, Vienna, Austria) will be started in women with serum E2 concentrations <200 pmol/l and no follicles >15 mm in diameter or ovarian cysts on ultrasonographic examination. The initial r-hFSH dose will be 250 IU s.c. daily for 5 days, after which the dose will be increased to a maximum of 450 IU per day using a step-up protocol with steps of 50 IU/day.
  Interventions: Drug: follicle stimulating hormone
- 2 (Active Comparator): No pituitary down-regulation will be performed. Treatment with r-hFSH (Gonal-F®, Serono Austria GmbH, Vienna, Austria) will be started in women with serum E2 concentrations <200 pmol/l and no follicles >15 mm in diameter or ovarian cysts on ultrasonographic examination. The r-hFSH dose will be 150 IU s.c. daily for 11 consecutive days.
  Interventions: Drug: follicle stimulating hormone

INTERVENTIONS:
Drug: follicle stimulating hormone — Pituitary down-regulation will be achieved using buserelin (Suprefact®, Hoechst, Frankfurt, Germany) at a fixed daily dose of 200 mg s.c., according to a long agonist protocol, starting on day 2 of the normal menstrual cycle. Treatment with r-hFSH (Gonal-F®, Serono Austria GmbH, Vienna, Austria) will be started in women with serum E2 concentrations <200 pmol/l and no follicles >15 mm in diameter or ovarian cysts on ultrasonographic examination. The initial r-hFSH dose will be 250 IU s.c. daily for 5 days, after which the dose will be increased to a maximum of 450 IU per day using a step-up protocol with steps of 50 IU/day.
  Other Names: buserelin, r-hFSH, r-hLH
  Arms: 1
Drug: follicle stimulating hormone — No pituitary down-regulation will be performed. Treatment with r-hFSH (Gonal-F®, Serono Austria GmbH, Vienna, Austria) will be started in women with serum E2 concentrations <200 pmol/l and no follicles >15 mm in diameter or ovarian cysts on ultrasonographic examination. The r-hFSH dose will be 150 IU s.c. daily for 11 consecutive days.
  Other Names: buserelin, r-hFSH, HCG
  Arms: 2

SUMMARY:
Available data from in vitro studies and clinical trials indicate that genetic factors play a significant role in the success of controlled ovarian stimulation (COS) prior to in vitro fertilization - embryo trandfer (IVF-ET). Women with the FSHR Ser680Asn Ser/Ser genotype make up between 13% and 26% of women undergoing IVF-ET and are characterised by higher basal FSH serum concentrations, the need for a higher amount of FSH for COS, and a higher risk of poor response to COS and cycle cancellation.

The investigators therefore intend to perform a study to investigate whether a dose-intensified COS protocol based on FSHR genotype status in women with the FSHR Ser680Asn Ser/Ser genotype is more effective than routine management in terms of

* the mean number of follicles
* the mean number of embryos
* the rate of poor responders
* the rate of women with cycle cancellations, and v) the clinical pregnancy rates.

Eligible women will be randomized to a stimulation protocol characterised by a longer duration and increased dosage of FSH stimulation (group A) or a standard stimulation protocol (group B).

DETAILED DESCRIPTION:
Women in group A will undergo controlled ovarian stimulation according to the following protocol:

Pituitary down-regulation will be achieved using buserelin (Suprefact®, Hoechst, Frankfurt, Germany) at a fixed daily dose of 200 mg s.c., according to a long agonist protocol, starting on day 2 of the normal menstrual cycle. Treatment with r-hFSH (Gonal-F®, Serono Austria GmbH, Vienna, Austria) will be started in women with serum E2 concentrations <200 pmol/l and no follicles >15 mm in diameter or ovarian cysts on ultrasonographic examination. The initial r-hFSH dose will be 250 IU s.c. daily for 5 days, after which the dose will be increased to a maximum of 450 IU per day using a step-up protocol with steps of 50 IU/day.

Once the leading follicle has reached a diameter of 14 mm, patients will receive r-hLH (lutropin alfa; Luveris®, Serono Austria GmbH, Vienna, Austria) at a dose of 75 IU s.c. for a maximum of 10 days. A dose of 75 IU LH per day was chosen based on findings from a controlled, prospective, dose-finding study in gonadotrophin-deficient women (WHO I classification) (7). Ovulation will be induced by administration of HCG (Profasi®, Serono Austria GmbH, Vienna, Austria), 10 000 IU i.m. or s.c., when at least two follicles have reached a diameter of >17 mm.

Oocyte retrieval will be performed by ultrasound-guided follicular aspiration techniques 34-38 h after administration of HCG. IVF will be performed according to standard practices at our institution. A maximum of three embryos will be transferred 48 h after oocyte retrieval (ESHRE Committee on Good Clinical and Laboratory Practice, 1995 ). Patients will receive micronized progesterone, 600 mg/day, by vaginal administration for at least the first 3 weeks of pregnancy, beginning on the day of embryo transfer.

Women in group B will undergo ovarian hyperstimulation according to the following protocol:

No pituitary down-regulation will be performed. Treatment with r-hFSH (Gonal-F®, Serono Austria GmbH, Vienna, Austria) will be started in women with serum E2 concentrations <200 pmol/l and no follicles >15 mm in diameter or ovarian cysts on ultrasonographic examination. The r-hFSH dose will be 150 IU s.c. daily for 11 consecutive days.

Once the leading follicle has reached a diameter of 14 mm, patients will receive r-hLH (lutropin alfa; Luveris®, Serono Austria GmbH, Vienna, Austria) at a dose of 75 IU s.c. for a maximum of 10 days. A dose of 75 IU LH per day was chosen based on findings from a controlled, prospective, dose-finding study in gonadotrophin-deficient women (WHO I classification) (European Recombinant Human LH Study Group, 1998 ). Ovulation will be induced by administration of HCG (Profasi®, Serono Austria GmbH, Vienna, Austria), 10 000 IU i.m. or s.c., when at least two follicles have reached a diameter of >17 mm.

Oocyte retrieval will be performed by ultrasound-guided follicular aspiration techniques 34-38 h after administration of HCG. IVF will be performed according to standard practices at our institution. A maximum of three embryos will be transferred 48 h after oocyte retrieval (ESHRE Committee on Good Clinical and Laboratory Practice, 1995 ). Patients will receive micronized progesterone, 600 mg/day, by vaginal administration for at least the first 3 weeks of pregnancy, beginning on the day of embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40
* Informed consent
* Indication for IVF-ET

Exclusion Criteria:

* Inability to understand written informed consent form
* Personal history of ovarian hyperstimulation syndrome

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 165 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | 3 months

SECONDARY OUTCOMES:
follicle count, cycle cancellation rate, poor responder rate | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Johannes C. Huber, MD, PhD, Study Director — Medical University of Vienna
Locations (1):
- University of Vienna, Vienna, Vienna, Austria